CLINICAL TRIAL: NCT06520384
Title: Comparison of Radiofrequency Applications and Alcoholic Neurolysis of Genicular Nerve for the Treatment of Knee Osteoarthritic Pain: A Randomized Trial
Brief Title: Radiofrequency Applications and Alcoholic Neurolysis of Genicular Nerve for the Treatment of Knee Osteoarthritic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR671/4/24
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Radiofrequency; Alcohol; Genicular Nerve; Knee Osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Radiofrequency group (Experimental): Patients will receive radiofrequency.
  Interventions: Device: Radiofrequency
- 30% alcohol group (Experimental): Patients will receive ultrasound-guided injection of each of the three genicular nerves with 0.5-0.75 ml of a solution containing 30% alcohol in 0.25% bupivacaine.
  Interventions: Drug: Alcohol 30%
- 50% alcohol group (Experimental): Patients will receive ultrasound-guided injection of each of the three genicular nerves with 0.5-0.75 ml of a solution containing 50% alcohol in 0.25% bupivacaine.
  Interventions: Drug: Alcohol 50%
- 70% alcohol group (Experimental): Patients will receive ultrasound-guided injection of each of the three genicular nerves with 0.5-0.75 ml of a solution containing 70% alcohol in 0.25% bupivacaine.
  Interventions: Drug: Alcohol 70%

INTERVENTIONS:
Device: Radiofrequency — Patients will receive radiofrequency.
  Arms: Radiofrequency group
Drug: Alcohol 30% — Patients will receive ultrasound-guided injection of each of the three genicular nerves with 0.5-0.75 ml of a solution containing 30% alcohol in 0.25% bupivacaine.
  Arms: 30% alcohol group
Drug: Alcohol 50% — Patients will receive ultrasound-guided injection of each of the three genicular nerves with 0.5-0.75 ml of a solution containing 50% alcohol in 0.25% bupivacaine.
  Arms: 50% alcohol group
Drug: Alcohol 70% — Patients will receive ultrasound-guided injection of each of the three genicular nerves with 0.5-0.75 ml of a solution containing 70% alcohol in 0.25% bupivacaine.
  Arms: 70% alcohol group

SUMMARY:
This study aims to investigate the efficacy of radiofrequency ablation and alcoholic neurolysis of genicular nerve on alleviating pain and improving the function of advanced knee osteoarthritis patients.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a major cause of pain and disability. Patients with moderate to severe knee OA often suffer from excruciating pain with chronic inflammation and reduced range of motion.

Conventional treatment of knee OA includes nonpharmacologic therapies and pharmacologic therapies. Analgesics, low-potency opioids, narcotic analgesics, and nonsteroidal anti-inflammatory drugs (NSAIDs) are commonly used in pharmacologic therapies.

Radiofrequency ablation (RFA) has been used for the treatment of chronic pain that has been unresponsive to conservative therapies. It acts by disrupting the transmission of pain signals using thermal lesion production to interrupt nociceptive signals.

The nerve block is conventionally performed by local anesthesia alone or in combination with corticosteroid. Nerve ablation causes iatrogenic neural degeneration aiming only for sensory or sympathetic denervation without motor deficits. The nerve ablation methods currently available are performed by either thermal ablation using RFA or chemical ablation using alcohol or phenol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Both sexes.
* Patients with knee osteoarthritis.
* Previous conservative treatments longer than 3 months.
* visual analog scale (VAS)≥ 4.
* Radiological osteoarthritis grades 3 and 4 according to the Kellgren-Lawrence grading system (0 = none, 1 = doubtful, 2 = minimal, 3 = moderate, and 4 = severe).

Exclusion Criteria:

* Patient refusal.
* History of knee surgery.
* Radiculopathy.
* Anticoagulant therapy.
* Injection with steroids or hyaluronic acids during the previous 3 months.
* Serious neurologic or psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Degree of knee pain | 6 months postoperative
  The degree of knee pain will be assessed using the visual analog scale (VAS). Each patient will obtain a score between 0 and 10 (Zero means no pain, and 10 means the worst pain). VAS will be assessed preoperative and postoperative 1, and 6 months

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores | 6 months postoperative
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): range from 0 to 96 (0 represents the best health status and 96 the worst possible status). The higher the score, the poorer the function. It will be assessed preoperative and postoperative 1, and 6 months.
Patient satisfaction | 6 months postoperative
  Degree of patient satisfaction will be assessed on a 5-point Likert scale Patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied ; 5, extremely satisfied).
Incidence of adverse events | 6 months postoperative
  Incidence of adverse events such as bleeding, neurological damage, infection, abnormal proprioception, numbness, paresthesia, and motor weakness will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.